CLINICAL TRIAL: NCT07119606
Title: Multicenter Study of Patients With SHANK3 Mutations: Identification of Genes Modificators in Phelan-McDermid Syndrome (EUQ13)
Acronym: EUQ13
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP231664; IDRCB: 2024-A02249-38 (Registry Identifier: IDRCB ANSM)
Record Dates: First submitted 2025-06-02; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-05

CONDITIONS: Genetic Disease
MeSH Terms: conditions — Genetic Diseases, Inborn | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHANK3 Mutation (Experimental)
  Interventions: Diagnostic Test: SHANK3 mutation

INTERVENTIONS:
Diagnostic Test: SHANK3 mutation — blood sampling for diagnostic test
  Other Names: blood sampling

SUMMARY:
Phelan-McDermid syndrome (PMS) is a neurodevelopmental disorder with extensive clinical and genetic heterogeneity that is still poorly understood. The phenotype includes hypotonia, delayed psychomotor development, intellectual disability of varying severity, and consistent language impairment ranging from delayed to absent speech. Autism spectrum disorders are present in 60-80% of patients, and other comorbidities may be present. The major candidate gene for PMS is SHANK3, which encodes a scaffolding protein in the dense postsynaptic region of glutamatergic synapses. Its loss of function is caused by deletions in the distal region of chromosome 22, 22q13.3, or by intragenic genomic variants. Several studies, including the one conducted by our team, have shown that part of the variability in the phenotype is related to the size of the 22q13.3 deletion. However, two patients with a deletion of similar size or an identical point variation in SHANK3 can have phenotypes of very variable severity.

The existence of additional genomic variants not identified by standard diagnostic techniques, particularly DNA chip chromosomal analysis (ACPA), which may act as modulating elements of the phenotype, has been suggested.

The limitations of the proposed studies are the highly heterogeneous genomic tools used (variable DNA chip design in terms of probe distribution and resolution) and the often imprecise phenotypes. Our study will bring together a large number of SPM patients (related to a 22q13.3 deletion or a variation of the SHANK3 gene) as well as their parents and possible relatives (first or second degree of the patient), very well phenotyped and explored by complete genome sequencing on the same sequencing platform.

DETAILED DESCRIPTION:
Phelan-McDermid syndrome (PMS) is a neurodevelopmental disorder (NDD) with a highly heterogeneous phenotype (Phelan & McDermid, 2011) characterized by hypotonia, delayed psychomotor development, intellectual disability of varying severity, and consistent language impairment ranging from simple delay to complete absence of language. Autism spectrum disorders are present in 60-80% of PMS patients, and other comorbidities are variably present (Kolevzon et al., 2014; Tabet et al., 2017). The major candidate gene for the syndrome is SHANK3, which encodes a scaffolding protein of the dense postsynaptic region of glutamatergic synapses, playing a fundamental role in the maintenance and function of these synapses. Loss of function of the SHANK3 gene can be caused by deletions in the distal region of chromosome 22, 22q13.3, or by intragenic genomic variants of the gene. SHANK3 proteins have several isoforms due to the presence of promoters and alternative splicing. Thus, an intragenic loss-of-function mutation at the beginning of the sequence will not have the same consequences as a mutation appearing at the end of the sequence. There is great heterogeneity, both clinical and genetic, among PMS patients.

A preliminary French study conducted by our team focused on the clinical and genetic analysis of 85 patients carrying CNV (Copy number variation, i.e. losses or gains of genetic material) covering the SHANK3 gene, identified by chromosomal microarray analysis (ACPA) as part of the genetic diagnosis of their pathology. This observational study confirmed that the size of the 22q13 deletion contributed to the variability of the syndrome, but also identified regions associated with particular phenotypic traits, as well as the presence of associated CNVs that could act as a phenotype-modifying factor (Tabet et al., 2017). The limitations of this study were 1- the diversity of the genetic tools used (highly variable resolution and design of DNA chips), 2- the very incomplete phenotyping of the included patients and 3- the absence of genomic sequencing data, thus excluding patients carrying intragenic SHANK3 variants and all other possible sequence variations (SNVs). In order to confirm the presence and possible impact of additional genomic variants (both CNVs and SNVs) in the variability of the syndrome, a very high resolution whole genome study (WGS) is necessary on a larger cohort of clinically well-phenotyped patients.

Furthermore, there is currently no specific treatment for PMS. Patients benefit from multidisciplinary care. A cellular model generated by Professor Benchoua's team has provided treatment prospects. Indeed, a screening of more than 200 molecules applied to neurons derived from induced pluripotent stem cells from patients carrying a truncating variant in SHANK3 showed that lithium increased SHANK3 expression and acted on various neuronal alterations. In particular, lithium re-increased the number of SHANK3-positive synapses as well as the frequency and intensity of spontaneous calcium oscillations. On a human scale, this study suggests that lithium can improve the neurodevelopmental disorder of patients. (Darville et al, 2016). Based on this work, a therapeutic trial is currently being implemented at Robert Debré Hospital (https://ichgcp.net/fr/clinical-trials-registry/NCT04623398). It includes patients carrying truncating variants in SHANK3 or small deletions involving SHANK3 and carriers of autism spectrum disorders. Studying the genome of the patients included in this study would also make it possible to establish correlations between the response to lithium and the genetic profile of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with Phelan-McDermid syndrome as part of the etiological assessment of a neurodevelopmental disorder, regardless of age (and their parents, siblings, and grandparents).
* For patients: identification of a deletion affecting SHANK3 or a specific, deleterious genetic variation in SHANK3.
* Affiliation to a social security scheme or beneficiary.
* Signature of the project consent form by the participant (if an adult) or by both legal guardians (if the participant is a minor or an adult under guardianship).

Exclusion Criteria:

-

Ages: 3 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Better Understanding the Clinical Variability of the Phelan-McDermid Syndrome | 18 months
  * Through precise characterization of the variation affecting the SHANK3 gene: mutation type, location of the variant, impact on the protein, and the specific SHANK3 isoform involved.
  * By identifying additional genetic variations (outside of SHANK3) that may contribute to associated conditions such as epilepsy, cardiopathy, or gastrointestinal disorders.
  * In cases of 22q13.3 deletions that include SHANK3-and therefore lead to a neurodevelopmental disorder-when additional genes are also affected by the deletion, better understanding the contribution of each of these genes to the presence and severity of associated clinical features.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Claude TABET, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debré Hospital, Paris, Ap-hp / DRCI, France